CLINICAL TRIAL: NCT04758299
Title: At Home Self-testing Kits for SARS-CoV-2 (Severe Acute Respiratory Syndrome Coronavirus 2) : A Randomized Trial Assessing How Consumers Interpret and Act on Test Results
Brief Title: Understanding Communications Included With COVID-19 (Corona Virus Disease of 2019) Home Testing Kits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barry Dewitt (Other)
Collaborators: Dartmouth College (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Barry Dewitt, Postdoctoral Research Associate, Carnegie Mellon University
Organization: Carnegie Mellon University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY2020_501
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: COVID-19 Testing; Decision Making

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either information from the FDA authorized home test kit for what actions to take for a negative or positive COVID-19 test (usual care) or a decision science-based design of similar length (intervention).
  There are 4 groups (clinical scenarios) within each randomized arm (the scenarios are patient with no symptoms and no exposure; no symptoms and exposure; symptoms and no exposure; symptoms and exposure.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): information from an FDA authorized home test kit for what actions to take for a negative or positive COVID-19 test
- Decision science-based design (Experimental): Information from a decision science-based design (of similar length to the FDA authorized home test kit information) for what actions to take for a negative or positive COVID-19 test
  Interventions: Other: decision science-based design

INTERVENTIONS:
Other: decision science-based design — decision science-based design explaining actions to take for a negative or positive COVID-19 test
  Arms: Decision science-based design

SUMMARY:
To test competing sets of information for consumers on how to interpret hypothetical SARS-CoV-2 home test kit results and whether they report plans to take CDC-recommended actions to protect themselves and others given their test results and two critical aspects of their clinical context: symptoms, recent close exposures. Participants will be randomized to receive either information from the FDA authorized Ellume home test kit (the first kit authorized for over the counter use) for what actions to take for a negative or positive COVID-19 test (usual care) or a decision science-based design of similar length (intervention).

DETAILED DESCRIPTION:
To test competing sets of information for consumers on how to interpret hypothetical SARS-CoV-2 home test kit results and whether they report plans to take CDC [Centers for Disease Control]-recommended actions to protect themselves and others given their test results and two critical aspects of their clinical context: symptoms, recent close exposures. Participants will be randomized to receive either information from the FDA authorized Ellume home test kit (the first kit authorized for over the counter use) for what actions to take for a negative or positive COVID-19 test (usual care) or a decision science-based design of similar length (intervention).

Participants will be randomized to receive either information from the FDA authorized Ellume home test kit for what actions to take for a negative or positive COVID-19 test (usual care) or a decision science-based design of similar length (intervention). They will be given time to read the documents and the opportunity to download a full "instructions for use" document (the FDA authorized for the ELLUME test kit). They will then be randomized to one of four conditions, asking them to imagine a clinical context: a person with no symptoms and no close COVID-19 contact, no symptoms and close contact,

ELIGIBILITY:
Inclusion Criteria:

* Participants must be >18 years old, communicate in English, reside in the United States.

Exclusion Criteria:

* Respondents who complete the survey in under a minute.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2021-03-13 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
choice of action to take with negative test | day 1
  choice of actions consistent with CDC-recommendations (eg, isolate or not) for various clinical scenarios (eg, with/without known exposure, with/without symptoms)
  Which of the following are safe for Jamie to do over the next week about being around others? [safe, not safe]
  1. Take no additional precautions.
  2. Stay at home except to visit close family or friends. Take no additional precautions at home
  3. Stay at home except when going to the grocery store. Take no additional precautions at home
  4. Stay at home all the time, without exceptions. Take no additional precautions at home.
  5. Stay at home all the time, without exceptions and avoid contact with others, including others in the household

SECONDARY OUTCOMES:
Likelihood of COVID-19 infection (qualitative) | day 1
  Judgments about the likelihood of COVID-19 infection with a negative or positive test result
  How likely is it that Jamie is infected with COVID-19? (choose one)
  1. Definitely yes
  2. Very likely
  3. Likely
  4. Unlikely
  5. Very Unlikely
  6. Definitely not
Likelihood of COVID-19 infection (quantitative) | day 1
  Judgments about the likelihood of COVID-19 infection with a negative ot positive test result
  Response using a "slider" to capture numeric estimate
safe practices | day 1
  Change in intent to practice standard public health practices to reduce COVID-19 transmission (hand washing, social distancing, masks) - question asked before and after seeing test result
  What else do you think Jamie should do to protect himself and others from COVID-19? [choose: all of the time, most of the time, some of the time, a little of the time, none of the time] In general
  1. Wash hands often
  2. Avoid close contact with people who seem sick (e.g., cough, sneeze, fever)
  3. Stay home
     Outside your home
  4. Try to avoid crowds
  5. Wear a mask when around others
  6. Keep 6 feet from others
  7. Avoid contact with anyone
ease of use of information rating | day 1
  how easy/hard is it to use information about interpreting test results
  How easy or difficult was it to read the information about interpreting the test result?" (check one)
  1. Very difficult
  2. Difficult
  3. Neutral
  4. Easy
  5. Very easy
usefulness of information rating | day 1
  how useful is the information about interpreting test results
  The information about interpreting the home test kit results was (check one)
  1. Extremely useful
  2. Useful
  3. Neutral
  4. Useless
  5. Completely useless
helpfulness of information for what to do given positive test result | day 1
  How helpful was the information for what to if test was positive
  The information helped me know what to do if test result is positive
  a. Strongly agree
  1. Agree
  2. Neutral
  3. Disagree
  4. Strongly disagree
helpfulness of information for what to do given negative test result | day 1
  How helpful was the information for what to if test was negative
  The information helped me know what to do if test result is negative
  a. Strongly agree
  1. Agree
  2. Neutral
  3. Disagree
  4. Strongly disagree
Assess effect of the FDA authorized description of test accuracy | day 1
  According to the test's FDA-authorized label, a clinical study conducted in the USA in 2020 showed that the test "correctly identified 96% of positive samples and 100% of negative samples in patients with symptoms. In people without symptoms the test correctly identified 91% of positive samples and 96% of negative samples."
  Based on this information, if Jamie has COVID now, what is the chance that the test will be wrong and say that he does not?
  RESPONSE (probability estimate) using slider

OTHER OUTCOMES:
ordering postest probability of infection | day 1
  correct ordering of posttest probability of infection risk (derived from qualitative and quantitative ratings)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Dewitt, Principal Investigator — Carnegie Mellon University; Steven Woloshin, MD, Principal Investigator — Dartmouth College; Tamar Krishnamurti, PhD, Principal Investigator — University of Pittsburgh; Baruch Fischhoff, PhD, Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woloshin S, Dewitt B, Krishnamurti T, Fischhoff B. Assessing How Consumers Interpret and Act on Results From At-Home COVID-19 Self-test Kits: A Randomized Clinical Trial. JAMA Intern Med. 2022 Mar 1;182(3):332-341. doi: 10.1001/jamainternmed.2021.8075. PMID 35099501